CLINICAL TRIAL: NCT02151253
Title: A Double-Blind, Placebo-Controlled, Cross-over Study of Armodafinil Treatment of Daytime Sleepiness Associated With Treated Nocturia
Brief Title: Cross-over Study of Armodafinil Treatment of Daytime Sleepiness Associated With Treated Nocturia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00028116
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Nocturia; Daytime Sleepiness
Keywords: Nocturia; Daytime sleepiness
MeSH Terms: conditions — Nocturia; Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armodafinil First, Then Placebo (Experimental): During double-blind treatment subjects took armodafinil for 4 weeks before crossing over to placebo for 4 weeks. Pill is taken once daily, before 8 am.
  Armodafinil/placebo was initiated at a dose of 50 mg (1 tablet) and titrated to 150 mg after 1 week on the basis of the investigator's and patient's perception of efficacy and side-effects. After two weeks the medication could be increased to 250 mg or reduced back to 50 mg based on the investigator's and patient's perception of efficacy/side-effects. No increases in dosage were allowed after week 2. The dosage was decreased at a week 3 phone call if indicated on the basis of side-effects.
  Interventions: Drug: Armodafinil; Drug: Placebo
- Placebo First, Then Armodafinil (Placebo Comparator): During double-blind treatment subjects took placebo for 4 weeks before crossing over to armodafinil for 4 weeks. Pill is taken once daily, before 8 am.
  Armodafinil/placebo was initiated at a dose of 50 mg (1 tablet) and titrated to 150 mg after 1 week on the basis of the investigator's and patient's perception of efficacy and side-effects. After two weeks the medication could be increased to 250 mg or reduced back to 50 mg based on the investigator's and patient's perception of efficacy/side-effects. No increases in dosage were allowed after week 2. The dosage was decreased at a week 3 phone call if indicated on the basis of side-effects.
  Interventions: Drug: Armodafinil; Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil — Armodafinil 50 - 250 mg pills Subjects took armodafinil once daily, before 8 am. Armodafinil was initiated at a dose of 50 mg (1 tablet) and titrated to 150 mg after 1 week on the basis of the investigator's and patient's perception of efficacy and side-effects. After two weeks the medication could be increased to 250 mg or reduced back to 50 mg based on the investigator's and patient's perception of efficacy/side-effects. No increases in dosage were allowed after week 2. The dosage was decreased at a week 3 phone call if indicated on the basis of side-effects.
Drug: Placebo — Subject given placebo tablets to match Armodafinil pills. Subjects took placebo once daily, before 8 am. Placebo was initiated as 1 tablet and titrated to 3 tablets after 1 week on the basis of the investigator's and patient's perception of efficacy and side-effects. After two weeks the medication could be increased to 5 tablets or reduced back to 1 tablet based on the investigator's and patient's perception of efficacy/side-effects. No increases in dosage were allowed after week 2. The dosage was decreased at a week 3 phone call if indicated on the basis of side-effects.

SUMMARY:
The objective of the study is to evaluate armodafinil as a wakefulness-promoting therapy as a means of improving residual daytime sleepiness in patients with treated nocturia.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving standard-of-care therapy for nocturia based on assessment by study physician
2. Evaluation by study physician indicates that the patient meets criteria for either overactive bladder diagnosis, or nocturnal polyuria diagnosis.
3. Mean number of nocturia episodes at least 2 per night based on day sleep/bladder diary
4. Epworth Sleepiness Scale Score of at least 10
5. Clinical Global Impression of Sleepiness at least Moderate
6. Age 18-90 years inclusive

Exclusion Criteria:

1. Medications affecting urinary or sleep-wake function other than therapy for OAB o or NP within 5 half-lives of baseline assessment
2. Sleep disorders other than nocturia based on history and screening assessment
3. Unstable medical or psychiatry conditions
4. Medical or psychiatric conditions affecting sleep/wake or urologic function
5. Apnea-Hypopnea Index (AHI) ≥ 15 on screening polysomnogram
6. Periodic Leg Movement Arousal Index (PLMAI) ≥ 15 on screening polysomnogram
7. History of substance abuse or dependence in the last year
8. Regular consumption of over 800 mg of caffeine use
9. Shift-work in the 3 months prior to or during the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-one individuals signed consent and were screened for entry into this study. Thirty of these subjects met the inclusion/exclusion criteria but only 28 subjects were randomized to the study. (2 subjects withdrew consent prior to randomization).
Period: Overall Study
Arm/Group | Armodafinil First, Then Placebo | Placebo First, Then Armodafinil
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 28
Age, Customized [Mean (Standard Deviation); unit: years]
  Between 18 and 90 | 54.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 17
  Caucasian | 9
  Asian | 1
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Epworth Sleepiness Scale [ESS]
Description: Epworth sleepiness scale (ESS) is measure of subjective sleepiness. Tendency to fall asleep in 8 situations. Total varies from zero to 24. A ESS of 10 or less is considered normal. Change is calculated as value at baseline minus value at week 4.
Time Frame: Baseline, Week 4 of each phase
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale | 9.03 (5.18) | 9.73 (4.43)

2. Secondary Outcome: Clinical Global Impressions, Change in Severity of Excessive Daytime Sleepiness (EDS)
Description: Scale consists of a 7 point likert rating scale where the anchors were 1= "normal"; 2= "borderline sleepiness"; 3= "mild sleepiness"; 4= "moderate sleepiness"; 5= "marked sleepiness"; 6= "severe sleepiness"; and 7= "among the most extremely sleepy individuals"
Time Frame: week 4, of each phase
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale | 2.58 (1.03) | 3.12 (0.82)

3. Secondary Outcome: Mean Number of Naps/Day
Description: measurements are for the preceding week
Time Frame: week 4 of each phase.
Measure: Mean (Standard Deviation); unit: naps per day
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 28 | 28
naps per day | 0.48 (0.71) | 0.73 (1.20)

4. Secondary Outcome: Mean Number of Minutes Napped Per Day Based on Sleep Diary
Description: measurements are for the preceding week
Time Frame: week 4 of each phase.
Measure: Mean (Standard Deviation); unit: minutes napped per day
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 28 | 28
minutes napped per day | 38.9 (65.1) | 40.0 (61.3)

5. Secondary Outcome: Mean Number of Nocturic Events (Episode of Urination Preceded and Followed by Sleep)
Description: Nocturic Events is defined as an episode of urination preceded and followed by sleep. Measurements are for the preceding week
Time Frame: week 4 of each phase.
Measure: Mean (Standard Deviation); unit: Nocturic Events
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 28 | 28
Nocturic Events | 1.6 (1.1) | 1.89 (1.1)

ADVERSE EVENTS:
Arm/Group | Armodafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 11/28 | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil (N=28) | Placebo (N=28)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anxiety/Jitteriness (Psychiatric disorders) | 4 | 3
insomnia (Psychiatric disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Dizziness (General disorders) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes